CLINICAL TRIAL: NCT05230706
Title: Application of a Light/Dark Cycle in Preterm Neonates and Its Association With Shorter In-hospital Stay
Brief Title: Light/Dark Cycle Promotes Weight Gain in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Universidad Autónoma Benito Juárez de Oaxaca (Other); Hospital General Dr. Aurelio Valdivieso (Other); Centro Medico Nacional La Raza, IMSS (Other); Hospital General Regional No. 1 IMSS (Other Government)
Responsible Party: Principal Investigator, Alberto Manuel Angeles Castellanos, Principal Investigator, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FOSISS-272596
Record Dates: First submitted 2022-01-26; First posted 2022-02-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Preterm Infants
Keywords: Circadian rhythms; Chronotherapy; Melatonin; Neonatology; Weight gain
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Intervention Model Description: Subjects randomized to the experimental group were allocated to alternating light/darkness conditions as follows: from 07:00 to 19:00 hours the subjects were kept under normal room light conditions; from 19:00 to 07:00 of the following day the conditions were modified by placing the patient under an acrylic cephalic helmet which exposed them to light at 25 lux for 12 hours every day. The control group was kept under normal room light conditions (CBL) 24 hours a day.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (CBL) (No Intervention): The control group was kept under normal room light conditions (CBL) 24 hours a day (level of illumination was 275.82±14 lux during the day and 145.28±14 lux at night).
- Experimental (LDC) (Experimental): The experimental group were allocated to alternating light/darkness conditions as follows: from 07:00 to 19:00 hours the subjects were kept under normal room light conditions; from 19:00 to 07:00 of the following day the conditions were modified by placing the patient under an acrylic cephalic helmet (length: 27 cm; width: 27 cm; height: 17.5 cm; opening: 17x12 cm). The helmet was covered with surgical cloth (green or blue) folded to 50x60cm rectangles, leaving the frontal part open in order to maintain an adequate air flow. This intervention exposed infants in the experimental group to light at 25 lux for 12 hours every day, while during daytime the cloth was removed in order for study subjects to be exposed to regular room lighting.
  Interventions: Other: Cephalic helmet

INTERVENTIONS:
Other: Cephalic helmet — An acrylic headgear (length: 27 cm; width: 27 cm; height: 17.5 cm; opening: 17x12 cm) was placed on the patient's head. The helmet was covered with surgical cloth (green or blue) folded into 50x60cm rectangles, leaving the front part open to maintain adequate airflow.
  Arms: Experimental (LDC)

SUMMARY:
The study focuses on the use of light/dark alternation as chronotherapy to prevent deterioration and reduce morbidity and mortality in premature patients, as well as favoring circadian alteration after birth, which should lead premature infants to a better evolution in life. NICU.

With the hypothesis that exposure to light/dark cycles during hospitalization of preterm infants will decrease hospital stay. In addition, the light/dark cycle will allow a circadian organization of physiological variables such as salivary levels of cortisol and melatonin.

To identify the benefits of the light/dark cycle in the clinical maturation of preterm newborn patients and early hospital discharge in preterm newborns.

DETAILED DESCRIPTION:
Introduction Worldwide, Neonatal Intensive Care Units (NICU) are often maintained under 24-hour constant bright light (CBL) conditions, without significant variations in light intensity. As such, infants under these conditions are exposed to chaotic temporal signals, as opposed to predictable temporal signals, without cyclic variations in terms of sounds and light. Interestingly, the level of light to which premature infants are exposed represents an accessible environmental variable that can be easily controlled. Premature infants are generally maintained under CBL conditions for prolonged intervals, thus hampering their growth and development. CBL conditions can generate harmful effects to newborn eyes, and experimental studies have shown that newborn rats exposed to a CBL environment from the first day of birth develop damage in the cellular organization of the retina.

Previous studies have shown that a 12:12 hour light/darkness cycle (LDC) can promote an increase in infant sleep time, decrease feeding time and improve weight gain, compared with infants maintained in constant light or constant dark conditions. Further, evidence shows that infants exposed to a LDC since birth acquire circadian rhythmicity of activity/rest patterns as early as week 34 of life.

This study presents the results from a multicentric trial which sought to determine the benefits of implementing a LDC in the NICU of three different hospitals in Mexico. The primary endpoint was weight gain; secondary endpoints included early hospital discharge, salivary melatonin levels and the effect of reducing the intensity of nocturnal light in development of premature infants.

Methods Study Design and Participants This prospective, open-label, randomized multicentric clinical trial recruited patients in three different public-setting hospitals in Mexico between 2016 and 2020. Eligible patients were premature infants (gestational age <37 weeks) who were hospitalized in the low risk and high-risk neonatal units of participating institution, with a non-severe diagnosis for hospitalization, without concomitant illness, and classified as stable. Exclusion criteria included infants hospitalized with severe illness, congenital malformations, or important neurological diseases, while elimination criteria included infants initially classified as having a non-severe illness who progress to severe illness, infants who received intensive treatment for over a week due to medical complications (i.e. bacterial infections), as well as infants whose parents requested withdrawal from participating in the study. The parents or legal guardians of all included patients provided written informed consent to participate in this study. Participating institutions included Centro Medico Nacional "La Raza", Mexico City; Hospital General de Zona No.1 "Dr. Demetrio Mayoral Pardo" Oaxaca City, Oaxaca, Mexico (both hospitals from the public healthcare system "Mexican Institute for Social Security IMSS"), and General Hospital "Dr. Aurelio Valdivieso", Oaxaca City, Oaxaca, Mexico (from the public healthcare system of the Health Secretariat [SSA]). The study was approved by the scientific and bioethical committees of each participating institution (CMNR-No. 3504-35, HGZ 1 IMSS Oaxaca R-2001-2015-8, SSO-R. 023/2018 y UNAM-094/2014). The study was performed in accord with the declaration of Helsinki and the principles of good clinical practice. This study followed the Consolidated Standards of Reporting Trials (CONSORT) reporting guidelines.

Sample Size The sample size was calculated for a two-sample comparison, given an 80% sensitivity and a 60% specificity and with a confidence interval of 90%. A total of 150 patients per group was estimated, for a total sample size of 300 subjects.

Procedures All study procedures were performed following a predefined study protocol and a uniform sample processing plan. Data was registered using a unified registry form in all participating sites, and all analyses were centrally performed at the main investigation site. All included patients provided information regarding family and perinatal history.

Each NICU from the participating institutions was evaluated in order to measure the illumination level using a luxmeter (HER-410-Steren), in 4 specific areas during 6 different times of day to ascertain homogeneous lighting conditions throughout the centers. Subjects randomized to the experimental group were allocated to alternating light/darkness conditions as follows: from 07:00 to 19:00 hours the subjects were kept under normal room light conditions; from 19:00 to 07:00 of the following day the conditions were modified by placing the patient under an acrylic cephalic helmet (length: 27 cm; width: 27 cm; height: 17.5 cm; opening: 17x12 cm). The helmet was covered with surgical cloth (green or blue) folded to 50x60cm rectangles, leaving the frontal part open in order to maintain an adequate air flow. This intervention exposed infants in the experimental group to light at 25 lux for 12 hours every day, while during daytime the cloth was removed in order for study subjects to be exposed to regular room lighting. The control group was kept under normal room light conditions (CBL) 24 hours a day (level of illumination was 275.82±14 lux during the day and 145.28±14 lux at night). All included subjects were under 24-hour surveillance for the period spanning the length of their hospital stay by the NICU personnel at each participating institution. Infants were kept in individual incubators regulated to maintain a body temperature ranging from 36.5 °C -37 °C.

Both study groups were offered feeding every 3 hours (as per NICU guidelines and vital signs were recorded every 3 hours (cardiac and respiratory rate, temperature). Every infant underwent an 8-12 hour fast after birth for intestinal resting, thereafter enteral feeding began at a dose of 12.5 ml/kg of breast milk, which was increased every 12 hours until reaching a maximum of 200 ml/kg/day. Every included infant was orally fed, in case of abdominal distension or absence of peristalsis underwent a 24-hour maximum fast. Once the infants reached 1600 g body weight, breast feeding was indicated in order to prepare for discharge. The total caloric content among different hospitals was not standardized in this present study.

Among 20 randomly selected infants (10 randomized to BCL and 10 randomized to LDC) saliva samples were collected two times a day (08:00, 23:00) every day during the first 20 days of NICU stay in order to determine biomarkers. The salivary concentration of melatonin was determined using a standardized ELISA kit, following instructions by the manufacturer (IBL International GmbH Flughafenstr. Hamburg, Germany).

Other procedures performed included capillary blood glucose, administration of medication as prescribed by their primary care physician, and sample acquisition for laboratory testing pertaining each condition presented by infants included in this trial. All included patients were monitored four weeks post hospital discharge to evaluate development and growth at home, as well as their circadian activity/rest patterns.

Healthy premature infants were considered for discharge when participants presented an adequate growth curve and met established growth criteria, including the ability to maintain a stable body temperature in an open crib, ability to perform all feedings without respiratory distress, and a constant weight gain >2000g.

Statistical Analysis Continuous variables were summarized as arithmetic means with standard deviations or medians and ranges according to the data distribution assessed with the Kolmogorov-Smirnov test. For descriptive purposes, categorical variables were summarized as frequencies and percentages. Data pertaining to body weight gain, feeding and melatonin concentration were classified per study group and evaluated as repeated measures according to post-natal days. Comparisons among study groups were performed using a two-way ANOVA, followed by a TUKEY post-test analysis. A p-value <0.5 was considered statistically significant. The initial body weight, gestational week, and length of hospital stay were compared using a one-way ANOVA, a p-value <0.5 was considered statistically significant. All analyses were performed using the STATISTICA program (V10; StatSoft, Inc. 1993), while figures were constructed using the program Sigma Plot (V14; Systat Software, San Jose, CA).

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were premature infants (gestational age <37 weeks) who were hospitalized in the low risk and high-risk neonatal units of participating institution, with a non-severe diagnosis for hospitalization, without concomitant illness, and classified as stable.
* The parents or legal guardians of all included patients provided written informed consent to participate in this study.

Exclusion Criteria:

* Exclusion criteria included infants hospitalized with severe illness, congenital malformations, or important neurological diseases-
* Elimination criteria included infants initially classified as having a non-severe illness who progress to severe illness, infants who received intensive treatment for over a week due to medical complications (i.e. bacterial infections), as well as infants whose parents requested withdrawal from participating in the study.

Ages: 1 Week to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Weight gain | The body weight gain during the initial 29 days of hospitalization
  Was determined by daily weighting (08:00-09:00 hours of every morning) using a pediatric precision scale, the result was subtracted from the previous day registered weight in order to obtain the total daily weight gain.

SECONDARY OUTCOMES:
Early hospital discharge | through study completion, an average of 8 weeks
  Time elapsed between the admission of the newborn to the neonatal care unit and discharge home
Salivary melatonin levels | The first 20 days of NICU stay
  Saliva samples were collected two times a day (08:00, 23:00) every day

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Manuel Angeles Castellanos, Principal Investigator — Universidad Nacional Autonoma de Mexico

IPD SHARING:
Plan to Share IPD: Yes
All the IPD of the results that underlie the publication will be shared when requested to the person in charge, in the time that is specified.
Supporting Information: SAP, ICF, CSR
Time Frame: As of 6 months after publication
Access Criteria: All the IPD of the results can be requested directly from the person in charge of the study, complying with the established time

REFERENCES:
- [Background] Escobar C, Rojas-Granados A, Angeles-Castellanos M. Development of the circadian system and relevance of periodic signals for neonatal development. Handb Clin Neurol. 2021;179:249-258. doi: 10.1016/B978-0-12-819975-6.00015-7. PMID 34225966
- [Background] Vasquez-Ruiz S, Maya-Barrios JA, Torres-Narvaez P, Vega-Martinez BR, Rojas-Granados A, Escobar C, Angeles-Castellanos M. A light/dark cycle in the NICU accelerates body weight gain and shortens time to discharge in preterm infants. Early Hum Dev. 2014 Sep;90(9):535-40. doi: 10.1016/j.earlhumdev.2014.04.015. Epub 2014 May 13. PMID 24831970
- [Background] Rivkees SA. Developing circadian rhythmicity. Basic and clinical aspects. Pediatr Clin North Am. 1997 Apr;44(2):467-87. doi: 10.1016/s0031-3955(05)70486-7. PMID 9130930
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174
- [Derived] Sanchez-Sanchez M, Garcia TL, Heredia D, Resendiz I, Cruz L, Santiago J, Rojas-Granados A, Ubaldo-Reyes L, Perez-Campos-Mayoral L, Perez-Campos E, Vasquez GS, Moguel JM, Zarate R, Garcia O, Sanchez L, Torres F, Paz A, Elizarraras-Rivas J, Hernandez-Huerta MT, Angeles-Castellanos M. Effect of a light-darkness cycle on the body weight gain of preterm infants admitted to the neonatal intensive care unit. Sci Rep. 2022 Oct 20;12(1):17569. doi: 10.1038/s41598-022-22533-1. PMID 36266474